CLINICAL TRIAL: NCT02128542
Title: A Phase 4, Multicenter, Open Label Study to Investigate the Efficacy and Safety of an All Oral Combination of Sofosbuvir+Ribavirin in Genotype 2 HCV-infected U.S. Veterans With Cirrhosis VALOR-HCV: Veterans Affairs alL Oral Regimen of SOF+RBV in GT2 HCV
Brief Title: Efficacy and Safety of Sofosbuvir+Ribavirin in Genotype 2 HCV-infected U.S. Veterans With Cirrhosis
Acronym: VALOR-HCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-1379
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C Virus Infection
Keywords: Veterans HCV
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sofosbuvir+RBV 12 weeks (Experimental): Participants will receive sofosbuvir+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will examine the safety, tolerability, and antiviral efficacy of sofosbuvir (SOF)+ribavirin (RBV) in treatment-naive and treatment-experienced United States Veterans with compensated cirrhosis and genotype 2 HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Treatment-naive or treatment-experienced adult, U.S. Veteran
* Chronic genotype 2 (GT2) HCV infection Classified as:

  * Eligible for treatment with interferon (IFN)-based therapy
  * Ineligible for IFN treatment
  * Intolerant to IFN.
* Cirrhosis determination
* Laboratory parameters within prespecified ranges at screening:
* A negative serum pregnancy test is required for females of childbearing potential
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Lactating females must agree to discontinue nursing before study drug is administered.
* Males must agree to refrain from sperm donation from the date of screening until at least 7 months after the last dose of RBV, or 90 days after their last dose of study drug if not taking RBV.
* Must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.
* Must be of generally good health as determined by the Investigator.

Exclusion Criteria:

* Current participation in an interventional clinical trial.
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
* History of any other clinically significant chronic liver disease (e.g., hemochromatosis; Wilson's disease; α1-antitrypsin deficiency), except nonalcoholic steatohepatitis (NASH).
* Decompensated liver
* History of hemoglobinopathies
* Contraindication or hypersensitivity to RBV
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the participation for the full duration of the study, such that it is not in the best interest of the individual to participate.
* Clinically significant ECG abnormality at screening.
* History of solid organ transplantation.
* Presence of hepatocellular carcinoma (HCC) Malignancy within 5 years prior to screening, with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer and prostate cancer in remission). Individuals under evaluation for possible malignancy are not eligible.
* Prior treatment with an NS5B polymerase inhibitor.
* Chronic use of systemic immunosuppressive agents or immunomodulatory agents (e.g., prednisone equivalent > 10 mg/day).
* Concomitant disallowed as per the Sovaldi Packet Insert.
* Known hypersensitivity to the study drug, the metabolites, or formulation excipient.
* History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
* Use of any prohibited concomitant medications as described in the study protocol
* Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug.
* Male with pregnant female partner.
* In the judgment of the investigator any clinically-relevant drug or alcohol abuse within 12 months of screening that may interfere with treatment, assessment or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Rossaro, MD, Study Director — Gilead Sciences
Locations (17):
- United States (17):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - New Haven, Connecticut
  - Miami, Florida
  - Decatur, Georgia
  - Baltimore, Maryland
  - Kansas City, Missouri
  - Durham, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia

REFERENCES:
- [Result] Ho SB, Monto A, Peyton A, Kaplan DE, Byrne S, Moon S, Copans A, Rossaro L, Roy A, Le H, Dvory-Sobol H, Zhu Y, Brainard DM, Guyer W, Shaikh O, Fuchs M, Morgan TR; VALOR study team. Efficacy of Sofosbuvir Plus Ribavirin in Veterans With Hepatitis C Virus Genotype 2 Infection, Compensated Cirrhosis, and Multiple Comorbidities. Clin Gastroenterol Hepatol. 2017 Feb;15(2):282-288. doi: 10.1016/j.cgh.2016.05.024. Epub 2016 May 27. PMID 27237429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 15 study sites in the United States The first participant was screened on 04 June 2014. The last study visit occurred on 22 June 2015.
Pre-assignment Details: 113 participants were screened.
Groups:
- SOF+RBV 12 Weeks (TN): Treatment-naive (TN) participants received sofosbuvir (Sovaldi®; SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
- SOF+RBV 12 Weeks (TE): Treatment-experienced participants received sofosbuvir (Sovaldi®; SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
Period: Overall Study
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE)
Started | 47 | 19
Completed | 43 | 19
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: participants who received at least 1 dose of study drug
Groups:
- SOF+RBV 12 Weeks (TN): Treatment-naive participants received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
- SOF+RBV 12 Weeks (TE): Treatment-experienced participants received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE) | Total
Number analyzed (Participants) | 47 | 19 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (6.0) | 62 (5.4) | 63 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 47 | 19 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 8 | 2 | 10
  White | 37 | 17 | 54
  Hawaiian or Pacific Islander | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 19 | 66
IL28b Status [Number; unit: participants]
  CC | 25 | 8 | 33
  CT | 19 | 10 | 29
  TT | 3 | 1 | 4
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.89) | 6.6 (0.48) | 6.1 (0.87)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 21 | 2 | 23
  ≥ 800,000 IU/mL | 26 | 17 | 43
HCV Genotype [Number; unit: participants]
  Genotype 2 | 2 | 2 | 4
  Genotype 2b | 37 | 17 | 54
  Genotype 2a/2c | 8 | 0 | 8
Cirrhosis Status [Number; unit: participants]
  No | 0 | 0 | 0
  Yes | 47 | 19 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled into the study and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 47 | 19
Percentage of participants | 76.6 [62.0 to 87.7] | 84.2 [60.4 to 96.6]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Groups:
- SOF+RBV 12 Weeks (All): All participants received SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
Arm/Group | SOF+RBV 12 Weeks (All)
Number analyzed (Participants) | 66
Percentage of participants | 4.5

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 47 | 19
percentage of participants | 78.7 [64.3 to 89.3] | 89.5 [66.9 to 98.7]

4. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough was defined as either:
  * HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment
  * HCV RNA ≥ LLOQ at the last available on-treatment measurement with no subsequent follow-up values
Time Frame: Up to Posttreatment Weak 12
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 47 | 19
Percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period after having achieved HCV RNA < LLOQ at end of treatment.
Time Frame: Up to Posttreatment Week 12
Population: Participants in the Full Analysis Set with available data were analyzed
  .
Measure: Number; unit: Percentage of participants
Groups:
- SOF+RBV 12 Weeks (TN); SOF+RBV 12 Weeks (TE): SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
Arm/Group | SOF+RBV 12 Weeks (TN) | SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 46 | 19
Percentage of participants | 17.4 | 15.8

6. Secondary Outcome: Number of Participants With Nonstructural Protein 5B (NS5B) Nucleoside Inhibitor (NI) Resistance-Associated Variants (RAVs) and RBV RAVs at Pretreatment and Posttreatment
Description: Deep sequencing of the HCV NS5B gene was attempted for all participants who had virologic failure at pretreatment and posttreatment time points if the level of HCV RNA in the plasma sample was ≥ 1000 IU/L.
Time Frame: Pretreatment and Posttreatment Week 12
Population: Participants who relapsed and qualified for sequencing analysis were analyzed.
Measure: Number; unit: participants
Arm/Group | SOF+RBV 12 Weeks (All)
Number analyzed (Participants) | 10
participants
  NS5B NI RAV Pretreatment | 2
  NS5B NI RAV Posttreatment | 5
  NS5B RBV RAV Pretreatment | 0
  NS5B RBV RAV Posttreatment | 0

ADVERSE EVENTS:
Time Frame: Up to12 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- SOF+RBV 12 Weeks (All Participants): SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks.
Arm/Group | SOF+RBV 12 Weeks (All Participants)
Serious Adverse Events (participants affected / at risk) | 8/66
Other Adverse Events (participants affected / at risk) | 45/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (All Participants) (N=66)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Drug withdrawal convulsions (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (All Participants) (N=66)
Anaemia (Blood and lymphatic system disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 11
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years